CLINICAL TRIAL: NCT00482703
Title: A Randomized, Multicenter, Open-label Phase II Study of Dasatinib (BMS-354825) Administered Orally at a Dose of 50mg Twice Daily or 100mg Once Daily in Subjects With Chronic Phase Philadelphia Chromosome Positive Chronic Myeloid Leukemia Who Are Resistant or Intolerant to Imatinib
Brief Title: A Study of Dasatinib in Chronic Phase Philadelphia Chromosome Positive Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-138
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-11

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: Imatinib resistant or intolerant chronic phase CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Dasatinib
- B (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: Dasatinib — tablets, Oral, 100 mg, once daily
  Other Names: Sprycel; BMS-354825
  Arms: A
Drug: dasatinib — tablets, Oral, 50 mg, twice daily
  Other Names: Sprycel; BMS-354825
  Arms: B

SUMMARY:
The objective is to evaluate the cytogenetic response to Dasatinib (BMS-354825) administered for 24 weeks in subjects with Imatinib resistant or intolerant chronic phase chronic myeloid leukemia (CML) once daily (QD) or twice daily. (BID)

ELIGIBILITY:
Inclusion Criteria:

* Philadelphia chromosome positive or bcr-abl gene positive Chronic phase Chronic Myelogenous Leukemia (CML) subjects must have primary or acquired resistance to Imatinib mesylate or have intolerance of imatinib mesylate
* Performance status (general conditions) specified by the Eastern Cooperative Oncology Group: 0-2
* Men and women, ages 20 to 75
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 3 months after the study in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Subjects who are eligible and willing to undergo transplantation at pre-study
* Women who are pregnant or breastfeeding
* Uncontrolled or significant cardiovascular disease
* History of significant bleeding disorder unrelated to CML
* Adequate hepatic function
* Adequate renal function
* Medication that increases bleeding risk
* Medication that changes heart rhythms
* Subjects who are compulsory detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Japan (9):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Nishinomiya-Shi, Hyōgo
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Isehara-Shi, Kanagawa
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Shibuya-Ku, Tokyo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib 100 mg Once-daily (QD) Starting Dose: Starting dose of 100 mg QD oral continuous daily dosing of Dasatinib (BMS-354825) for 24 weeks. One dose escalation allowed for nonresponding participants; dose reduction mandated according to the observed toxicity.
- Dasatinib 50 mg Twice-daily (BID) Starting Dose: Starting dose of 50 mg BID oral continuous daily dosing of Dasatinib (BMS-354825) for 24 weeks. One dose escalation allowed for nonresponding participants; dose reduction mandated according to the observed toxicity.
Period: Overall Study
Arm/Group | Dasatinib 100 mg Once-daily (QD) Starting Dose | Dasatinib 50 mg Twice-daily (BID) Starting Dose
Started | 11 (number enrolled, randomized and treated) | 12 (number enrolled, randomized and treated)
Completed | 10 | 12
Not Completed | 1 | 0
Not completed — Poor compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100 mg Once-daily (QD) Starting Dose | Dasatinib 50 mg Twice-daily (BID) Starting Dose | Total
Number analyzed (Participants) | 11 | 12 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (14.2) | 49.9 (16.0) | 49.3 (14.8)
Age, Customized [Number; unit: participants]
  <65 years | 9 | 10 | 19
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Japan | 11 | 12 | 23
Eastern Cooperative Oncology Group Performace Status (ECOG-PS) [Number; unit: participants] — ECOG PS scale is a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale=0-5, with 0=fully active, 1=restricted in physically strenuous activity but ambulatory, 2=ambulatory and capable of all selfcare but unable to work, 3= limited selfcare ability and confined to bed/chair >50% of waking hours, 4=completely disabled and no selfcare ability and confined to bed/chair, and 5=death
  participants
    Status=0 | 11 | 12 | 23
    Status=1 | 0 | 0 | 0
    Status=2 | 0 | 0 | 0
    Status=3 | 0 | 0 | 0
    Status=4 | 0 | 0 | 0
    Status=5 | 0 | 0 | 0
Imatinib Status [Number; unit: participants] — Resistance to Imatinib=Previously treated with imatinib at a dose of ≥ 400 mg/day AND developed progressive disease while receiving imatinib at that dose. Intolerance to Imatinib=development of a Grade ≥3 toxicity considered at least possibly related to imatinib at a dose of ≤400 mg/day which led to discontinuation of therapy.
  participants
    Imatinib-resistant | 7 | 7 | 14
    Imatinib-intolerant | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cytogenetic Response in Imatinib-Intolerant and Imatinib-Resistant Participants at Week 24
Description: Cytogenetic responses (CyR) are based on the percentage of Philadelphia-positive (Ph+) metaphases among at least 20 metaphase cells in each bone marrow (BM) sample. The criteria for cytogenetic responses are as follows. Best CyR is defined as the best response obtained at any time during the study. Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), and Partial Cytogenetic Response (PCyR; 1 - 35 Ph+ Cells in Metaphase in BM).
Time Frame: Week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dasatinib 100 mg QD Starting Dose Cohort: All participants treated with a starting Dasatinib (BMS-354825) dose of 100 mg QD oral continuous daily dosing (CCD) for 24 weeks.
- Dasatinib 100 mg QD Starting Dose - Imatinib-resistant: Imatinib-resistant participants treated with a starting Dasatinib (BMS-354825) dose of 100 mg QD oral continuous daily dosing (CCD) for 24 weeks.
- Dasatinib 100 mg QD Starting Dose - Imatinib-intolerant: Imatinib-intolerant participants treated with a starting Dasatinib (BMS-354825) dose of 100 mg QD oral continuous daily dosing (CCD) for 24 weeks.
- Dasatinib 50 mg BID Starting Dose Cohort: All participants treated with a starting Dasatinib (BMS-354825) dose of 50 mg BID oral continuous daily dosing (CCD) for 24 weeks.
- Dasatinib 50 mg BID Starting Dose - Imatinib-resistant: Imatinib-resistant participants treated with a starting Dasatinib (BMS-354825) dose of 50 mg BID oral continuous daily dosing (CCD) for 24 weeks.
- Dasatinib 50 mg BID Starting Dose - Imatinib-intolerant: Imatinib-intolerant participants treated with a starting Dasatinib (BMS-354825) dose of 50 mg BID oral continuous daily dosing (CCD) for 24 weeks.
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 100 mg QD Starting Dose - Imatinib-resistant | Dasatinib 100 mg QD Starting Dose - Imatinib-intolerant | Dasatinib 50 mg BID Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose - Imatinib-resistant | Dasatinib 50 mg BID Starting Dose - Imatinib-intolerant
Number analyzed (Participants) | 11 | 7 | 4 | 12 | 7 | 5
percentage of participants
  MCyR | 45 [16.7 to 76.6] | 29 [3.7 to 71.0] | 75 [19.4 to 99.4] | 92 [61.5 to 99.8] | 86 [42.1 to 99.6] | 100 [47.8 to 100.0]
  CCyR | 27 [6.0 to 61.0] | 14 [0.4 to 57.9] | 50 [6.8 to 93.2] | 58 [27.7 to 84.8] | 43 [9.9 to 81.6] | 80 [28.4 to 99.5]

2. Secondary Outcome: Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuations, and Deaths During Treatment
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Throughout study period to last observation. Dosing period=6 months; if beneficial, medication may continue in the extension period (ending in January 2009). Last observation=30 days past last dosing day or the discontinuation day.
Population: All treated participants
Measure: Number; unit: participants
Groups:
- Dasatinib 100 mg QD Starting Dose Cohort: All participants treated with a starting dose of Dasatinib (BMS-354825) 100 mg QD oral continuous daily dosing (CCD) for 24 weeks.
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 11 | 12
participants
  AEs (symptoms/signs and laboratory abnormalities) | 11 | 12
  SAEs (symptoms/signs and laboratory abnormalities) | 4 | 6
  Deaths | 0 | 0
  AEs that led to discontinuation | 0 | 0

3. Secondary Outcome: Complete Hematologic Response (CHR) in Imatinib-Intolerant and Imatinib-Resistant Participants at Week 24
Description: CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm³; no blasts or promyelocytes in peripheral blood; < 5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils < 20%; no extramedullary involvement. A confirmed CHR (cCHR) is obtained when all above criteria are maintained for at least 28 days after they are first met. All hematologic responses can begin only 14 days after the dosing start date.
Time Frame: Week 24
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 100 mg QD Starting Dose - Imatinib-resistant | Dasatinib 100 mg QD Starting Dose - Imatinib-intolerant | Dasatinib 50 mg BID Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose - Imatinib-resistant | Dasatinib 50 mg BID Starting Dose - Imatinib-intolerant
Number analyzed (Participants) | 11 | 7 | 4 | 12 | 7 | 5
percentage of participants | 91 [58.7 to 99.8] | 86 [42.1 to 99.6] | 100 [39.8 to 100.0] | 83 [51.6 to 97.9] | 86 [42.1 to 99.6] | 80 [28.4 to 99.5]

4. Secondary Outcome: Time to Major Cytogenetic Response (MCyR)
Description: Time to MCyR is defined as the time from first dose of Dasatinib (BMS-354825) until the first day criteria for CCyR or PCyR, whichever occurs first, are first met. MCyR = a complete and a partial cytogenetic response (CyR), based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow sample. Percentage of Ph+ Cells in Metaphase in bone marrow: Complete Cytogenetic Response (CCyR) = 0; Partial Cytogenetic Response (PCyR) 1 - 35
Time Frame: time from first dose of Dasatinib (BMS-354825) until the first day criteria for CCyR or PCyR, whichever occurs first, are first met
Population: Treated participants - responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 6 | 11
months | 5.5 [5.3 to 5.6] | 4.2 [2.8 to 5.2]

5. Secondary Outcome: Pharmacokinetics of Dasatinib (BMS-354825) as Characterized by Population Pharmacokinetics
Description: Blood sample collection for pharmacokinetic (PK) analysis that will contribute to PK modeling.
Time Frame: Six or more peripheral blood samples were collected at any visit after Day 7, pre-dose and 5 - 8 hours after dose administration.
Population: Blood samples were collected for PK to be included in separate population PK analyses. No study specific PK analyses were planned for this report.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of MCyR
Description: The duration of MCyR will be measured from the first day all criteria are met for CCyR or PCyR until the date of progressed disease (PD) or death. Subjects who neither progress nor die will be censored on the date of their last cytogenetic assessment.MCyR = a complete and a partial cytogenetic response (CyR), based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow sample. Percentage of Philadelphia-positive (Ph+) Cells in Metaphase in bone marrow: Complete Cytogenetic Response (CCyR) = 0; Partial Cytogenetic Response (PCyR) 1 - 35
Time Frame: from the first day all criteria are met for CCyR or PCyR until the date of progressed disease (PD) or death
Population: Median duration was not reached at the time of this report; see Outcome Measure 14 for corresponding life table.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to CHR
Description: Time to CHR = time from first dose of Dasatinib until the first day CHR criteria are met (provided subjects achieved a cCHR). CHR=all of the following criteria: white blood cell count ≤ upper limit of normal; platelets <450,000/mm³; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils <20%; no extramedullary involvement. A confirmed CHR (cCHR) is obtained when all above criteria are maintained for at least 28 days after they are first met. All hematologic responses can begin only 14 days after the dosing start date.
Time Frame: time from first dose of Dasatinib (BMS-354825) until the first day CHR criteria are met
Population: Treated participants - responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 10 | 10
months | 1.0 [0.5 to 1.1] | 0.6 [0.5 to 0.9]

8. Secondary Outcome: Duration of CHR
Description: The duration of CHR were measured from the first day all criteria were first met for CHR (provided subjects achieved a cCHR), until the date PD is first reported or until death. Subjects who neither progress nor die were censored on the date of their last hematologic assessment.
Time Frame: measured from the first day all criteria were first met for CHR (provided subjects achieved a cCHR), until the date PD is first reported or until death
Population: Median duration of CHR was not reach at the time of this report. See corresponding life table presented in Outcome Measure 15.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progressed disease=achieving a CHR & subsequently no longer meeting criteria consistently over a consecutive 2-week period after starting maximum dose; no CHR after receiving maximum dose & increase in white blood cell count (doubling of count from lowest value to >20,000/mm3 or an increase by >50,000/mm3 on 2 assessments done ≥2 weeks apart); meeting the criteria of accelerated or blastic phase chronic myeloid leukemia at any time; having an MCyR & subsequently no longer meeting the criteria for MCyR after starting maximum dose; or having a >=30% absolute increase in number of Ph+ metaphases.
Time Frame: as for outcome 4
Population: Median months of progression-free survival was not reached at the time of this report. See corresponding life table in Outcome Measure 16.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Expression of BCR-ABL Gene Mutations of RNA (mRNA)
Description: Number of participants with positive (>= 2.0 log copies/mg) and negative (<2.0 log copies/mg) expression of mRNA at Baseline and at end of study.
Time Frame: Baseline and at the end of long term extension period (The enrollment period was followed by an extension period until the launch of dasatinib in Japan, January 2009.)
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 11 | 12
participants
  Positive at Baseline | 11 | 11
  Negative at Baseline | 0 | 1
  Positive at End-of-Study | 8 | 3
  Negative at End-of-Study | 3 | 9

11. Secondary Outcome: Mutational Spectrum of BCR-ABL
Description: Number of participants with a particular BCR-ABL mutation at Baseline and End-of-Study.
Time Frame: as for outcome 10
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 11 | 12
participants
  G250E mutation at Baseline | 1 | 3
  G250E mutation at End-of-Study | 1 | 0
  F317L mutation at Baseline | 0 | 0
  F317L mutation at End-of-Study | 1 | 0
  T315I mutation at Baseline | 0 | 1
  T315I mutation at End-of-Study | 0 | 1

12. Secondary Outcome: Cytogenetic Response in Imatinib-Intolerant and Imatinib-Resistant Participants at End of Study
Description: Cytogenetic response (CyR) as reflected in the major cytogenetic response was determined by bone marrow (BM) aspirates and are based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each BM sample. Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR; 0 Ph+ Cells in Metaphase in BM), or Partial Cytogenetic Response (PCyR; 1 - 35 Ph+ Cells in Metaphase in BM).
Time Frame: as for outcome 10
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 11 | 12
percentage of participants
  MCyR | 55 [23.4 to 83.3] | 92 [61.5 to 99.8]
  CCyR | 36 [10.9 to 69.2] | 67 [34.9 to 90.1]

13. Secondary Outcome: Hematologic Response in Imatinib-Intolerant and Imatinib-Resistant Participants at End of Study
Description: as for outcome 3
Time Frame: as for outcome 10
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 11 | 12
percentage of participants | 91 [58.7 to 99.8] | 83 [51.6 to 97.9]

14. Other Pre Specified Outcome: Number of Participants With Major Cytogenetic Response at Months 0 - 24 (Duration of MCyR Life Table)
Description: MCyR = a complete and a partial cytogenetic response (CyR), based on the percentage of Ph+ metaphases among at least 20 metaphase cells in each bone marrow sample. Percentage of Ph+ Cells in Metaphase in BM: Complete Cytogenetic Response (CCyR) = 0; Partial Cytogenetic Response (PCyR) 1 - 35
Time Frame: Months 0, 4, 8, 12, 16, 20, 24
Population: Treated participants. Median duration was not reached at the time of this report (see Outcome Measure 6)
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 6 | 11
participants
  Month 0 | 6 | 11
  Month 4 | 6 | 9
  Month 8 | 6 | 9
  Month 12 | 4 | 8
  Month 16 | 3 | 3
  Month 20 | 0 | 1
  Month 24 | 0 | 0

15. Other Pre Specified Outcome: Number of Participants With CHR at Months 0 - 24 (Duration of MCyR Life Table)
Description: as for outcome 3
Time Frame: Months 0, 4, 8, 12, 16, 20, 24
Population: Treated participants. Median duration was not reached at the time of this report (see Outcome Measure 7)
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 6 | 11
participants
  Month 0 | 10 | 10
  Month 4 | 9 | 10
  Month 8 | 9 | 8
  Month 12 | 9 | 8
  Month 16 | 8 | 7
  Month 20 | 4 | 4
  Month 24 | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Progression-Free Survival (PFS) at Months 0 - 24 (PFS Life Table)
Description: Progressed disease=achieving a CHR and subsequently no longer meeting criteria consistently over a consecutive 2-week period after starting maximum dose; no CHR after receiving maximum dose and an increase in white blood cell count (doubling of the count from lowest value to >20,000/mm3 or an increase by >50,000/mm3 on 2 assessments done at least 2 weeks apart); meeting the criteria of accelerated or blastic phase CML at any time; having an MCyR and subsequently no longer meeting the criteria for MCyR after starting maximum dose; or having a >=30% absolute increase in number of Ph+ metaphases.
Time Frame: Months 0, 4, 8, 12, 16, 20, 24
Population: Treated participants. Median duration was not reached at the time of this report (see Outcome Measure 7)
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD Starting Dose Cohort | Dasatinib 50 mg BID Starting Dose Cohort
Number analyzed (Participants) | 6 | 11
participants
  Month 0 | 11 | 12
  Month 4 | 11 | 12
  Month 8 | 9 | 10
  Month 12 | 9 | 10
  Month 16 | 9 | 10
  Month 20 | 7 | 7
  Month 24 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dasatinib 100 mg Once-daily (QD) Starting Dose | Dasatinib 50 mg Twice-daily (BID) Starting Dose | Total
Serious Adverse Events (participants affected / at risk) | 4/11 | 6/12 | 10/23
Other Adverse Events (participants affected / at risk) | 11/11 | 12/12 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg Once-daily (QD) Starting Dose (N=11) | Dasatinib 50 mg Twice-daily (BID) Starting Dose (N=12) | Total (N=23)
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg Once-daily (QD) Starting Dose (N=11) | Dasatinib 50 mg Twice-daily (BID) Starting Dose (N=12) | Total (N=23)
Anaemia (Blood and lymphatic system disorders) | 6 | 6 | 12
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2 | 3
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 3 | 1 | 4
Cataract (Eye disorders) | 2 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1
Retinopathy (Eye disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 9
Constipation (Gastrointestinal disorders) | 1 | 5 | 6
Dental caries (Gastrointestinal disorders) | 3 | 1 | 4
Gastritis (Gastrointestinal disorders) | 4 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Oedema mouth (Gastrointestinal disorders) | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Gastric dysplasia (Gastrointestinal disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 6
Oedema peripheral (General disorders) | 2 | 2 | 4
Malaise (General disorders) | 2 | 1 | 3
Chest pain (General disorders) | 1 | 1 | 2
Face oedema (General disorders) | 0 | 2 | 2
Oedema (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 1 | 0 | 1
Feeling abnormal (General disorders) | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 7 | 10 | 17
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Platelet count decreased (Investigations) | 8 | 7 | 15
Neutrophil count decreased (Investigations) | 7 | 7 | 14
White blood cell count decreased (Investigations) | 5 | 7 | 12
Alanine aminotransferase increased (Investigations) | 3 | 6 | 9
Lymphocyte count decreased (Investigations) | 5 | 4 | 9
Blood creatine phosphokinase increased (Investigations) | 1 | 5 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 5 | 5
Blood phosphorus decreased (Investigations) | 3 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 4
Blood albumin decreased (Investigations) | 3 | 1 | 4
Blood creatinine increased (Investigations) | 3 | 1 | 4
Red blood cell count decreased (Investigations) | 1 | 3 | 4
Blood sodium decreased (Investigations) | 2 | 1 | 3
Haemoglobin decreased (Investigations) | 1 | 2 | 3
Liver function test abnormal (Investigations) | 0 | 3 | 3
Weight decreased (Investigations) | 1 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 3
Blood potassium decreased (Investigations) | 1 | 1 | 2
Blood urea increased (Investigations) | 2 | 0 | 2
Blood uric acid increased (Investigations) | 1 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 2
Weight increased (Investigations) | 1 | 1 | 2
Protein urine present (Investigations) | 1 | 1 | 2
Blood calcium decreased (Investigations) | 1 | 0 | 1
Blood fibrinogen increased (Investigations) | 1 | 0 | 1
Blood folate decreased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 1
Lymphocyte count increased (Investigations) | 1 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 1
Protein total increased (Investigations) | 0 | 1 | 1
Vitamin B12 decreased (Investigations) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 3 | 5
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Apathy (Psychiatric disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 9 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Skin depigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 3
Hypotension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.